CLINICAL TRIAL: NCT03360812
Title: Online Randomised Controlled Trial to Improve Clinical Estimates of Survival (ORaClES)
Brief Title: ORaClES: A Trial to Improve Prognostication
Acronym: ORaClES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Brunel University (Other); Imperial College London (Other); Marie Curie Hospice, Belfast (Other); Hull York Medical School (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 17/0650
Record Dates: First submitted 2017-11-23; First posted 2017-12-04 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Terminal Illness
Keywords: Medical Students; Education; Prognosis; Online training resource

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention is an online training resource to improve the recognition of imminent death in palliative care patients. The intervention should take approximately 15 minutes to complete. During this time, the participants who are in the intervention arm will be shown the results of a previous study which identified how expert palliative care doctors recognise imminently dying palliative care patients. The intervention will be implemented via the website, immediately after participants have completed the first set of vignettes.
  Interventions: Other: Online training resource
- Control group (No Intervention): The participants assigned to the control group will not receive this additional information and will simply be informed that they are approximately half way through the task and will be asked to continue on to the next set of vignettes.

INTERVENTIONS:
Other: Online training resource — Please see information included in the description of the intervention group.
  Arms: Intervention group

SUMMARY:
This study evaluates whether an online training resource can improve the performance of medical students in recognising imminently dying palliative care patients.

DETAILED DESCRIPTION:
Clinicians are routinely asked to provide survival estimates for palliative care patients, but recognition of imminent death (last 72 hours of life) is often inaccurate. We developed an online training resource, based on a previous study that identified the symptoms or signs that were most influential in forming expert palliative care doctors' prognostic decisions about imminent death.

This double-blind randomised controlled trial will evaluate the effectiveness of this online training resource in improving the performance of medical students in recognising imminently dying palliative care patients.

Participants are asked to visit the study website and review three series of vignettes describing patients referred to palliative care. For each vignette, participants are asked to provide an estimate (0-100%) about the probability that the patient will die in the next 72 hours. After the first series of vignettes, students randomised to the intervention arm are given access to an online training resource showing how experts weighted the relative importance of symptoms and signs. All participants are asked to complete a second series of vignettes. After two weeks, all participants are asked to return to the website and complete a third series of vignettes to assess if any effect has been maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Enrolled on a registered medical course within the United Kingdom
3. In the penultimate or final year of medical school
4. Sufficient English language proficiency
5. Willing and able to provide consent as indicated by taking part in the online survey

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-08-12 (Actual)

PRIMARY OUTCOMES:
Survival estimates - immediate effect | Second series of vignettes, taking into account the estimates from the first series. Students can participate at their convenience and will have a four week window to complete the first and second series of vignettes.
  The primary outcome will be a continuous survival estimate provided from the students for the second series of vignettes; ranging from 0-100%.

SECONDARY OUTCOMES:
Survival estimates - follow-up | Third series of vignettes, taking into account the estimates from previous series. Two weeks after completing the first and second series of vignettes, students will be asked to complete a third series of vignettes within a four week window.
  Survival estimates provided from the students at the two week follow-up; ranging from 0-100%.
Cue weighting | Change over time including all three series of vignettes. Students are given a four week window to complete the first and second series of vignettes. After two weeks, they will be asked to complete a third series of vignettes within a four week window.
  Cue weighting of the individual students as compared to the experts; that is the coefficient of each factor as part of their "judgement policy".
Level of expertise | Change over time including all three series of vignettes. Students are given a four week window to complete the first and second series of vignettes. After two weeks, they will be asked to complete a third series of vignettes within a four week window.
  The level of expertise will be assessed with the Cochran-Weiss-Shanteau (CWS) score. This score details the level of ability to discriminate and the level of consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, PhD, MD, Principal Investigator — UCL
Locations (5):
- United Kingdom (5):
  - Brighton and Sussex Medical School, Brighton
  - Hull York Medical School, Hull
  - Imperial College London, London
  - St George's Medical School, London
  - UCL Medical School, London

IPD SHARING:
Plan to Share IPD: Yes
Data (suitably anonymised) may be shared with other research groups if a reasonable request is submitted to and agreed by the Chief Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the publication of results and will be archived securely by the Chief Investigator for a minimum of 20 years from the declaration of end of trial.
Access Criteria: The data will be shared upon reasonable request.

REFERENCES:
- [Background] Oostendorp L, White N, Harries P, Yardley S, Tomlinson C, Ricciardi F, Gokalp H, Stone P. Protocol for the ORaClES study: an online randomised controlled trial to improve clinical estimates of survival using a training resource for medical students. BMJ Open. 2019 Mar 3;9(3):e025265. doi: 10.1136/bmjopen-2018-025265. PMID 30833321
- [Background] White N, Oostendorp LJ, Tomlinson C, Yardley S, Ricciardi F, Gokalp H, Minton O, Boland JW, Clark B, Harries P, Stone P. Online training improves medical students' ability to recognise when a person is dying: The ORaClES randomised controlled trial. Palliat Med. 2020 Jan;34(1):134-144. doi: 10.1177/0269216319880767. Epub 2019 Nov 14. PMID 31722611

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03360812/SAP_000.pdf